CLINICAL TRIAL: NCT03686553
Title: St. Barbara Specialised Regional Hospital No. 5: Surveillance of Healthcare-Associated Infections
Status: Completed | Type: Observational
Sponsor: Polskie Towarzystwo Zakażeń Szpitalnych (Other)
Responsible Party: Sponsor
Other Study IDs: PTZS
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Surgical Site Infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infected, with SSI: patients with SSI
  Interventions: Other: laboratory-based data collection
- non-infected: patients without SSI
  Interventions: Other: laboratory-based data collection

INTERVENTIONS:
Other: laboratory-based data collection — laboratory-based surveillance of SSI

SUMMARY:
Retrospective laboratory-based data collection study of surgical site infections: Surveillance of Healthcare-Associated Infections in Orthopaedic and Trauma Surgery Unit in Sosnowiec, Poland;

ELIGIBILITY:
Inclusion Criteria:

* patient being treated in the Department and Clinic of Orthopaedic and Trauma Surgery, St. Barbara Specialised Regional Hospital No. 5, Sosnowiec
* patients undergoing surgery in studied unit

Exclusion Criteria:

* under 18 years of age
* surgery of a different type than orthopedics
* non-surgical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing surgery in the Orthopaedic and Trauma Surgery Unit in Sosnowiec, Poland
Sampling Method: Probability Sample
Enrollment: 5239 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
surgical site infection incidence rate | The follow-up period was 30 days for the superficial SSI's, and 90 days for deep or organ/space infections following arthroplasties
  the cumulative incidence of surgical site infection (SSI) was calculated by dividing the number of SSI cases by the number of patients undergoing surgery and multiplying by 100

IPD SHARING:
Plan to Share IPD: No